CLINICAL TRIAL: NCT06902480
Title: Assessing Choline Bioavailability and Metabolism From a New Dairy Ingredient for Post-Menopausal Women
Brief Title: Dairy Choline Bioavailability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-1661; A074000 (Other: UW Madison); CALS/FOOD SCIENCE (Other: UW Madison); Protocol Version 8/21/25 (Other: UW Madison)
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Post-menopausal Women; Post-menopausal Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey Protein Phospholipid Concentrate (WPPC) (Experimental): Participants will drink a chocolate-flavored drink with WPPC added
  Interventions: Dietary Supplement: WPPC
- Pasteurized whole egg powder (Experimental): Participants will drink a chocolate-flavored drink with egg powder added
  Interventions: Dietary Supplement: Whole egg powder

INTERVENTIONS:
Dietary Supplement: WPPC — A chocolate-flavored drink with WPPC added
  Arms: Whey Protein Phospholipid Concentrate (WPPC)
Dietary Supplement: Whole egg powder — A chocolate-flavored drink with whole egg powder added
  Arms: Pasteurized whole egg powder

SUMMARY:
The goal of this clinical trial is to find out if dairy is a good source of choline compared to eggs. The main questions it aims to answer are:

* How the body uses choline; and,
* What effect WPPC has on choline metabolism.

Researchers will compare Whey Protein Phospholipid Concentrate (WPPC) to whole egg powder to see if WPPC is as effective as eggs.

Participants will drink a chocolate-flavored drink mixed with either WPPC or whole egg powder.

DETAILED DESCRIPTION:
This study is intended to evaluate the bioavailability and metabolism of choline in WPPC compared to the most commonly -used food for bioavailable choline, whole egg. The intent of the evaluation is to improve the knowledge of how WPPC contributes to the nutritional needs and health of postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 51 and 70
* Is currently post-menopausal (Post-menopausal is a term used to describe the time in a woman's life after she has gone through menopause. This usually happens between the ages of 45 and 55. Menopause is when a woman's menstrual periods stop permanently (at least 12 months))
* Not allergic to the intervention foods and allergens that are related to the production of intervention foods (e.g. dairy products, egg, fish, peanut, shellfish, soy, tree nuts, wheat, crustaceans, gluten, mollusks, mustard, sesame seeds.)
* Had stable body weight (± 5%) for the past 6 months
* Free from cancer
* Did not have weight loss surgery, colon surgery
* Do not have chronic kidney diseases
* Do not have malabsorption towards fat and dairy products
* Willing to complete health surveys
* Willing to complete two 4-day food diaries
* Willing to consume the intervention beverages
* Willing to provide blood, urine, fecal samples at baseline and after 10 days of intervention

Exclusion Criteria:

* On weight loss/weight gain diets
* Diagnosed with fat malabsorption
* Undergoing weight loss surgery
* Diagnosed with chronic kidney diseases
* Allergic to the intervention foods and allergens that are related to the production of intervention foods (e.g. dairy products, egg, chocolate, fish, peanut, shellfish, soy, tree nuts, wheat, crustaceans, gluten, mollusks, mustard, sesame seeds, banana, strawberry, raspberry, blackberry, blueberry.)
* Regularly using antibiotics or probiotics or prebiotics
* Regularly using Orlistat or Cetilistat
* Regularly using laxatives
* Undergoing hormone replacement therapy, or receiving hormones in any forms
* Unable to avoid strenuous exercise during the study (>4 h intense exercise per day)

Ages: 51 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in circulating choline | Baseline to 10 days
  Circulating choline will be measured by UHPLC-HRMS/MS

SECONDARY OUTCOMES:
Change in co-factors in circulating choline | Baseline to 10 days
  Co-factors in the circulation will be measured by ultrahigh performance liquid chromatography coupled with high resolution tandem mass spectrometry (UHPLC-HRMS/MS).
Change in high-sensitivity C-reactive protein (hs-CRP) | Baseline to 10 days
  Safety biomarker Hs-CRP will be measured using immunoturbidimetry.
Change in circulating choline metabolites | Baseline to 10 days
  Metabolites will be measured by UHPLC-HRMS/MS.
Change in 8-hydroxydeoxyguanosine | Baseline to 10 days
  The safety biomarker 8-hydroxydeoxyguanosine (8-OHDG) will be measured using enzyme-linked immunosorbent assay (ELISA).
Change in aspartate transaminase | Baseline to 10 days
  Aspartate transaminase (AST) will be measured using kinetic methods.
Change in alanine transaminase (ALT) | Baseline to 10 days
  Alanine transaminase will be measured using kinetic methods.
Change in creatinine | Baseline to 10 days
  Creatinine will be measured using kinetic methods

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Bolling, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share the individual participant data collected during the trial after deidentification. Deidentified data will be stored and shared with DryAd and in accordance with all applicable regulations.
Time Frame: Anticipated data availability will be immediately following publication. No end date.
Access Criteria: Data will be shared with DryAd. The data generated in this study will be housed in DryAd.
URL: https://datadryad.org/